CLINICAL TRIAL: NCT04204252
Title: Prospective Phase 3 Multi-center 2-Year Placebo Controlled Double Blind Study to Evaluate the Efficacy and Safety of Kamada-AAT for Inhalation 80 mg/Day in Alpha-1 Antitrypsin Deficiency With Moderate and Severe Airflow Limitation Followed by a 2-Year Open Label Extension
Brief Title: Phase III, Efficacy and Safety of "Kamada-AAT for Inhalation"
Acronym: InnovAATe
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kamada-AAT (inhaled) 008
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: Alpha 1 Antitrypsin; Inhaled Alpha 1 Antitrypsin; Nebulizer
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin; Inhalation

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized for 2 years of double-blind treatment with AAT for Inhalation 80 mg/d or placebo, followed by an additional 2 years of open label treatment with AAT for inhalation 80 mg/L. Participants will be followed up for safety for 24 weeks following the end of study treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled AAT (Active Comparator): Daily inhalation of 80 mg/day "Kamada-AAT for Inhalation" for 104 weeks
  Interventions: Drug: Alpha 1-Antitrypsin
- Placebo (Placebo Comparator): Daily inhalation of a solution of NaCl in phosphate buffer solution with 0.01% TWEEN-80
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alpha 1-Antitrypsin — Kamada's alpha 1-antitrypsin product given by inhalation using the eFlow® electronic nebulizer manufactured by PARI Pharma GmbH
  Other Names: Kamada alpha 1-antitrypsin for inhalation
  Arms: Inhaled AAT
Drug: Placebo — Preparation of NaCl in phosphate buffer solution with 0.01% TWEEN-80
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if AAT for inhalation, at a dose of 80 mg/day can slow the progression of lung disease in people who have lung disease caused by severe genetic deficiency in Alpha 1 Antitrypsin (AATD).

The main question it aims to answer is:

• Can daily treatment with Kamada AAT for inhalation at a dose of 80 mg/day prevent or slow lung function worsening ? Lung function will be measured by spirometry.

Other questions it aims to answer are:

* Can daily treatment with Kamada AAT for inhalation at a dose of 80 mg/day prevent or slow lung density loss ? Lung density will be measured by a CT scan.
* Can daily treatment with Kamada AAT for inhalation at a dose of 80 mg/day prevent or slow lung disease from worsening ? Lung disease will be measured using spirometry, lung volume, gas diffusion, six minute walk test, quality of life questionaires and biomarkers.
* What medical problems do participants have when taking AAT for inhalation 80 mg/day daily ? Researchers will compare AAT for inhalation to a placebo (a look-alike substance that contains no drug) to see if AAT for inhalation works to treat AAT-deficiency related lung disease. Study participants will receive either AAT for inhalation or placebo for the first two years of the study. During the third and fourth years of the study all participants will receive AAT for inhalation regardless of which drug they received during the first two years.

Participants will:

* Inhale the study drug every day
* Clean and disinfect the nebulizer every day
* Document daily symptoms and study drug use in an electronic diary
* Visit the clinic for tests and assessments. There are 11 clinic visits during the first two years of the study and 5-6 clinic visits during the third and fourth year, combined. After treatment ends, participants will visit the clinic 3 times in half a year.

DETAILED DESCRIPTION:
Individuals with a genetic deficiency of alpha-1-antitrypsin (AATD) are at a significantly increased risk (80-100%) of developing lung disease (emphysema or COPD). This study is designed to administer a solution of AAT by nebulizer so that patients can inhale the drug instead of requiring infusions as in current treatment. A significant advantage of inhalation is that the AAT is directly transferred to the lungs, which is the site most in need of the protein. Previous results show that in addition to the added convenience, treatment restores normal levels of active AAT to the lung. To date, more than 220 participants have completed clinical trials with AAT for inhalation for several diseases.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of severe AAT deficiency, i.e. patients with either Pi(ZZ), Pi(Z/Null), or Pi(Null/Null) genotypes.
2. Serum AAT levels ≤ 11 µM at screening.
3. Lung disease with clinical evidence of airflow limitation (post bronchodilator FEV1/SVC≤70%) at screening.
4. 40% ≤ FEV1 ≤ 80% of predicted post-bronchodilator at screening.
5. Patients who are either naïve or washed out of any AAT treatment for at least 8 weeks prior to randomization.
6. Age between 18 to 65 years inclusive at screening.
7. Able to read and sign informed consent and willing to participate in the study.
8. Males or non-pregnant, non-lactating females whose screening pregnancy test is negative, who are willing to use contraceptive methods for the duration of the study, or who are postmenopausal, or surgically sterilized.
9. Study medication use for at least 20 out of the 28 days of run-in, as recorded in the study nebulization PARI Track data.
10. Demonstrated ability to complete eDiary for at least 20 out of the first 28 days of run-in.

Exclusion Criteria

1. Immunoglobulin A (IgA) absolute deficiency defined as serum IgA levels < 0.05 g/L.
2. History of life-threatening transfusion reaction(s), allergy, anaphylactic reaction, or systemic response to human plasma-derived products.
3. Two or more moderate or any severe exacerbation(s) within the year prior to baseline.
4. A moderate exacerbation within 6 weeks prior to baseline.
5. Use of oral or parenteral glucocorticoids in doses above 10 mg of prednisone daily or equivalent generics (substance and dose).
6. Clinically significant inter-current illnesses (except for respiratory or liver disease secondary to AAT deficiency), including: cardiac, hepatic, renal, endocrine, neurological, hematological, neoplastic, immunological, skeletal, or other. Patients might be included after consultation with the treating physician and the sponsor if, in the opinion of the Investigator, their condition will not interfere with the safety, compliance or other aspects of this study.
7. Hospitalization for any cause during the 6 weeks prior to screening.
8. History of lung or liver transplant.
9. On any thoracic or hepatic surgery waiting list.
10. Any lung surgery within the past two years (including bronchoscopic lung volume reduction).
11. Any smoking within the year prior to screening.
12. Evidence of alcohol abuse or history of alcohol abuse, or use of illegal drugs and/or abuse of legally prescribed drugs in the last 5 years prior to screening.
13. Acute or chronic hepatitis (hepatitis A, hepatitis B, hepatitis C), or positive human immunodeficiency virus (HIV) serology.
14. Signs of significant abnormalities in serum hematology, serum chemistry, serum inflammatory / immunogenic markers and urinalysis per investigator judgment, taking into considerations the potential effects of the AAT deficiency.
15. Signs of significant abnormalities in ECG per investigator judgment at screening.
16. Presence of psychiatric/ mental disorder or any other medical disorder that might impair the patient's ability to give informed consent or to comply with the requirements of the study protocol. If, in the opinion of the Investigator, the condition will not interfere with the compliance or other aspects of this study, the patient might be included after consultation with the treating physician and the sponsor.
17. Participation in another clinical trial involving investigational medication or interventional treatment within 30 days and/or last dose 5 half-lives prior to screening visit.
18. Inability to attend scheduled clinic visits and/or comply with study protocol.
19. Any other factor that, in the opinion of the investigator, would prevent the patient from complying with the requirements of the protocol.

Additional eligibility criteria apply for the open label extension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
FEV1 post bronchodilator | 104 weeks
  Change from baseline in post bronchodilator FEV1 at 104 weeks

SECONDARY OUTCOMES:
CT densitometry whole-lung 15th percentile lung density (PD15) at total lung capacity (TLC). | 104 weeks
  Change from baseline over 104 weeks of treatment in CT densitometry whole-lung 15th percentile lung density (PD15) at total lung capacity (TLC).
FEV1 % of predicted | 104 weeks
  Change from baseline over 104 weeks of treatment in FEV1 % of predicted
FEV1/FVC % | 104 weeks
  Change from baseline over 104 weeks of treatment in FEV1/FVC %
Exacerbations | 104 weeks
  Annual rate of exacerbations by severity and duration
6 minute walk test | 104 weeks
  Change from Baseline in the distance walked in six minutes

OTHER OUTCOMES:
TEAEs | 130 weeks
  Rate and severity of adverse events during treatment emergent adverse events (TEAEs), adverse events of special interest (AESIs) and serious adverse events (SAEs) during treatment and follow-up period [Safety Outcome]
PiM | 130 weeks
  Plasma M-type AAT specific (PiM) levels evaluated as function of exposure time, antibody response (positive vs. negative), and antibody titers. [Safety Outcome]
ADA/nADA | 130 weeks
  Rate and titers of binding and neutralizing AAT antibodies (ADA/nADA) in plasma [Safety Outcome]
ECG | 130 weeks
  Electrocardiogram [Safety Outcome] will be classified as normal or abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stolk, Prof, Principal Investigator — LUMC
Locations (9):
- University Hospital (UZ) Leuven, Leuven, Belgium
- Tays Central Hospital, Tampere, Finland
- Beaumont Hospital, Dublin, Ireland
- Netherlands (2):
  - Leiden University Medical Center (LUMC), Leiden, ZA
  - Canisius Wilhelmina Hospital (CWZ), Nijmegen
- Skåne University Hospital, Malmo, Sweden
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kappe NN, Alagem N, Tov N, Stolk J. Governmental Non-Pharmaceutical Interventions during the COVID-19 Pandemic and the COPD Exacerbation and Respiratory Infection Rate in Patients with Alpha-1 Antitrypsin Deficiency. COPD. 2023 Dec;20(1):292-297. doi: 10.1080/15412555.2023.2249108. PMID 37665565